CLINICAL TRIAL: NCT06526923
Title: A Single Ascending Dose, Phase 1/2 Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of SP-101 Via Nebulizer for the Treatment of Cystic Fibrosis (CF)
Brief Title: A Phase 1/2 Trial of SP-101 for the Treatment of Cystic Fibrosis (CF)
Acronym: SAAVe
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spirovant Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CFAAV-001
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
Keywords: gene therapy; SP-101; AAV; doxorubicin; inhaled; augmenter
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Aspiration | interventions — EGFR inhibitor SP101; Doxorubicin

STUDY DESIGN:
Intervention Model Description: Single ascending dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Cohort 1 (Experimental): Single inhalational administration of SP-101 and doxorubicin Dose 1
  Interventions: Combination Product: SP-101 and doxorubicin Cohort 1
- Cohort 2 (Experimental): Single inhalational administration of SP-101 and doxorubicin Dose 2
  Interventions: Combination Product: SP-101 and doxorubicin Cohort 2
- Dose Expansion (Experimental): Single inhalational administration of SP-101 and doxorubicin Selected Dose
  Interventions: Combination Product: SP-101 and doxorubicin Cohort 1; Combination Product: SP-101 and doxorubicin Cohort 2

INTERVENTIONS:
Combination Product: SP-101 and doxorubicin Cohort 1 — Single inhaled dose of SP-101 and doxorubicin Dose 1
  Other Names: SP-101; doxorubicin
  Arms: Cohort 1; Dose Expansion
Combination Product: SP-101 and doxorubicin Cohort 2 — Single inhaled dose of SP-101 and doxorubicin Dose 2
  Other Names: SP-101; doxorubicin
  Arms: Cohort 2; Dose Expansion

SUMMARY:
This is a Phase 1/2 multicenter, open-label, single dose trial of SP-101 investigational gene therapy in adults with CF who are ineligible for or intolerant to CFTR modulator therapy.

DETAILED DESCRIPTION:
This multi-center study is a first-in-human, single ascending dose, Phase 1/2 trial to evaluate the safety, pharmacokinetics, and pharmacodynamics of various dose levels in people with CF who are ineligible or intolerant to CFTR modulator therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 to 65 years at Screening Visit, inclusive
2. Diagnosis of CF
3. ppFEV1 value between 50-100% (inclusive)
4. Resting oxygen saturation ≥94% on room air by pulse oximetry 5 . Clinically stable CF disease as assessed by the Investigator and not requiring any new class of interventional treatment within the last 3 months prior to Screening

Exclusion Criteria:

1. Any change in established pulmonary treatment (including antibiotics) within 28 days prior to Screening Visit. However, inhaled beta-agonists can be included within 2 weeks prior to Screening Visit.
2. Clinically significant episode of hemoptysis (>50 mL or ¼ cup or 10 teaspoons per day) within 12 weeks prior to dosing with study drug on Day 1
3. Lung infection with Mycobacterium abscessus associated with a more rapid decline in pulmonary status
4. Currently receiving treatment for active lung infection with Burkholderia cenocepacia or Burkholderia dolosa
5. History of solid organ or hematological transplantation
6. History of clinically significant cirrhosis with or without portal hypertension
7. History of pulmonary hypertension
8. History of cardiotoxicity, a history of known coronary artery disease, and/or existing cardiomyopathy
9. Current active fungal infection (not just a positive culture), acute blood, lung, or bladder infection, clinically significant hepatic or renal dysfunction, and/or viral infection (including human immunodeficiency virus or hepatitis virus B or C) requiring the initiation of new therapy within 30 days prior to Screening
10. History of allergic bronchopulmonary aspergillosis (ABPA)
11. Uncontrolled diabetes mellitus, as evidenced by hemoglobin A1c >9% at Screening
12. Clinically significant laboratory abnormalities at Screening
13. Subjects with any medical condition or abnormal laboratory result that, in the opinion of the Investigator, will interfere with the safe completion of the study
14. Subjects who received any investigational products within 30 days (or 5 therapeutic half-lives, whichever is longer) prior to Screening
15. Subjects who have previously received any gene therapy agent
16. Subjects with known sensitivity to SP-101, doxorubicin or its excipients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 52 weeks
  Safety and tolerability of SP-101 following a single inhalation dose, as assessed by incidence and severity of treatment emergent adverse events, serious adverse events, and dose limiting toxicities, including clinically significant changes from baseline to scheduled time points in safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lee, MPH, Study Director — Spirovant Sciences
Locations (4):
- United States (4):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - Hospital at University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Excoffon KJDA, Smith MD, Falese L, Schulingkamp R, Lin S, Mahankali M, Narayan PKL, Glatfelter MR, Limberis MP, Yuen E, Kolbeck R. Inhalation of SP-101 Followed by Inhaled Doxorubicin Results in Robust and Durable hCFTRDeltaR Transgene Expression in the Airways of Wild-Type and Cystic Fibrosis Ferrets. Hum Gene Ther. 2024 Sep;35(17-18):710-725. doi: 10.1089/hum.2024.064. Epub 2024 Sep 4. PMID 39155828
- [Result] Excoffon KJDA, Lin S, Narayan PKL, Sitaraman S, Jimah AM, Fallon TT, James ML, Glatfelter MR, Limberis MP, Smith MD, Guffanti G, Kolbeck R. SP-101, A Novel Adeno-Associated Virus Gene Therapy for the Treatment of Cystic Fibrosis, Mediates Functional Correction of Primary Human Airway Epithelia From Donors with Cystic Fibrosis. Hum Gene Ther. 2024 Sep;35(17-18):695-709. doi: 10.1089/hum.2024.063. Epub 2024 Aug 29. PMID 39155805